CLINICAL TRIAL: NCT05948358
Title: The Menstrual Distress Questionnaire (MEDI-Q) Reliability and Validity of the Turkish Version
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Nurcan Contarli, Principal Investigator, Karabuk University
Other Study IDs: Menstrual Distress
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Menstruation Disturbances
MeSH Terms: conditions — Menstruation Disturbances

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Females: 18 Years to 45 Years (Adult )
  Interventions: Other: Menstrual Distress Questionnaire

INTERVENTIONS:
Other: Menstrual Distress Questionnaire — The Menstrual Distress Questionnaire (MEDI-Q) is a new tool originally developed in Italian that comprehensively evaluates menstrual-related distress.

SUMMARY:
Menstruation is a process in which metabolic and hormonal changes occur periodically every month to maintain reproductive functions in women. This cycle, which continues from menarche to menopause, repeats approximately every 28 days and lasts 3-7 days (1). The menstrual cycle is divided into three phases, the follicular phase, the ovulation phase, and the luteal phase, in which the levels of estrogen and progesterone hormones change (2,3). In this cycle, which is regulated by the hormones released from the pituitary, hypothalamus and ovary, changes occur not only in the genital organs, but also in the nervous system, cardiovascular system, respiratory system, musculoskeletal system and metabolic functions (4). Responses to these changes, which cause physiological stress in the organism in women, are perceived in different degrees. The presence of recurrent abnormal bleeding or excessive pain may be a sign of various menstrual disorders (5). Evaluation of menstrual problems that negatively affect women's mood, social and work life is clinically important (6,7).

The scale, called Menstrual Distress Questionnaire (MEDI-Q), was developed by Vannuccini et al. (2021), it is a tool that comprehensively evaluates menstrual problems (8). MEDI-Q assesses the effects of menstrual symptoms on quality of life, recreational activities, work and social relationships. It consists of 25 items covering different areas of menstruation-related symptoms such as pain, discomfort, psychological and cognitive changes, and gastrointestinal disturbances. The level of distress caused by each symptom is assessed in the menstrual cycle phases, taking into account not only its impact on functionality and quality of life, but also its frequency. MEDI-Q is a scale with good test-retest reliability and internal consistency (Cronbach's = 0.85) (8,9). The scale provides a total score (MEDI-Q Total Score) and three subscales that assess general menstrual distress. Subscales; the number of distressing symptoms (MS) during menstruation, the mean level of distress related to menstrual symptoms (MSD), and the Menstrual Specificity Index (MESI) (8,9), which measures the proportion of symptoms at which distress exacerbates during the menstrual phase.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* 18-35 years old
* Volunteer
* Native speaker Turkish

Exclusion Criteria:

* Pregnancy or breastfeeding
* Having a mental health problem

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female university students between the ages of 18 and 45 who is native Turkish speaker
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
The Menstrual Distress Questionnaire (MEDI-Q) | 10 minutes
  The Menstrual Distress Questionnaire (MEDI-Q) is a new tool originally developed in Italian that comprehensively evaluates menstrual-related distress.

IPD SHARING:
Plan to Share IPD: No